CLINICAL TRIAL: NCT07310173
Title: Phase IIb, Randomized, Active-Controlled, Parallel-Group, Multicenter Clinical Study to Evaluate the Efficacy and Safety of AST-3424 in Patients With AKR1C3-High Expressing Advanced Hepatocellular Carcinoma Who Progressed After Systemic Therapy With Immune Checkpoint Inhibitors
Brief Title: Phase IIb Study of AST-3424 in Patients With AKR1C3-high Expressing Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSE001-Ⅱ-01
Record Dates: First submitted 2025-12-10; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AST3424, 4mg/m^2 (Experimental)
  Interventions: Drug: AST-3424
- AST3424, 6mg/m^2 (Experimental)
  Interventions: Drug: AST-3424
- regorafenib (Active Comparator)
  Interventions: Drug: Regorafenib Tablets

INTERVENTIONS:
Drug: AST-3424 — AST-3424 is administered via intravenous infusion on Day 1 and Day 8 of each 21-day treatment cycle
  Arms: AST3424, 4mg/m^2; AST3424, 6mg/m^2
Drug: Regorafenib Tablets — 160 mg orally, once daily for the first 21 days of each 28-day treatment cycle.
  Arms: regorafenib

SUMMARY:
The goal of this clinical trial is to learn if drug AST-3424 works to treat AKR1C3 high expressing advanced hepatocellular carcinoma after failure of systemic therapy with immune checkpoint inhibitors. The main question it aims to answer is:

Does AST-3424 prolong survival in patients with AKR1C3-high Expressing advanced Hepatocellular Carcinoma who have progressed after immune checkpoint inhibitors based therapies?

Researchers will compare AST-3424 to regorafenib (current optional therapy for target patients) to see if AST-3424 works.

Participants will:

Receive AST-3424 infusion on Day 1 and Day 8 of each 21-day treatment cycle or take regorafenib once a day on Day 1 -Day 21 of each 28-day treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed advanced hepatocellular carcinoma (HCC).
2. Documented disease progression confirmed by medical imaging after failure of prior systemic therapy regimens containing immune checkpoint inhibitors (ICIs).
3. Barcelona Clinic Liver Cancer (BCLC) stage B or C; ineligible for or refusing surgical resection or locoregional liver therapies (including transarterial intervention and ablation).
4. Child-Pugh class A or B liver function (score ≤ 7), with no history of hepatic encephalopathy.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
6. At least one measurable extracranial lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
7. Expected survival ≥ 3 months.
8. Availability of pathological tissue blocks or sections (including archived samples) for AKR1C3 expression and related biomarker analysis. Immunohistochemistry (IHC) results must confirm high expression of AKR1C3.
9. Adequate organ function.
10. For subjects positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb):

    HBV DNA level must be < 2000 IU/mL or 10⁴ copies/mL Subjects must be receiving anti-HBV therapy . This therapy must be maintained throughout the study period and for 6 months after the last dose of study drug.

    For subjects positive for HCV antibody, HCV-RNA level must be below the lower limit of detection (LLOD) of the study center.
11. Female subjects of childbearing potential must be non-lactating and have a negative pregnancy test result within 7 days prior to treatment initiation. A positive urine pregnancy test result must be confirmed by a serum pregnancy test.
12. Female and male subjects of childbearing potential must agree to use effective contraceptive measures from the time of study enrollment until 6 months after the last dose of study drug.
13. Subjects must voluntarily participate in the study, provide written informed consent after a full understanding of the study details, and have good compliance to cooperate with study treatment, observation, and follow-up procedures.

Exclusion Criteria:

1. Patients with intrahepatic cholangiocarcinoma, dual-phenotype hepatocellular carcinoma, fibrolamellar hepatocellular carcinoma, or carcinosarcoma.
2. Untreated active central nervous system (CNS) metastases. Subjects with CNS metastases who have received adequate treatment, achieved stable disease for at least 4 weeks confirmed by clinical examination and brain MRI during screening, require no steroid or anticonvulsant therapy, and present no clinical symptoms may be enrolled in the study.
3. A history of other malignant tumors within 2 years, except for adequately treated basal cell carcinoma of the skin, carcinoma in situ of the lung, breast, or other sites, or other tumors whose related treatments will not interfere with the safety or efficacy evaluation of the study drug.
4. A history of severe cardiovascular and cerebrovascular diseases.
5. Has received anti-tumor therapies including locoregional radiotherapy, chemotherapy, immunotherapy, or targeted therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose; for treatment with nitrosourea or mitomycin C, a 6-week washout period is required; for oral fluoropyrimidine drugs or small-molecule targeted therapy drugs, only a 2-week washout period is needed.
6. Has received major surgery other than diagnostic procedures or locoregional therapy targeting liver lesions within 4 weeks prior to the first dose.
7. Has received investigational drugs in other clinical trials within 4 weeks prior to the first dose.
8. All toxicities from prior anti-cancer therapies must have resolved to ≤ grade 1 at the start of study drug administration.
9. Moderate to large symptomatic pleural effusion, pericardial effusion, or ascites requiring thoracentesis/paracentesis or with a history of thoracentesis/paracentesis within 2 weeks prior to the start of study treatment. .
10. Need for concomitant use of strong CYP3A4 inhibitors or inducers during the study period.
11. Any severe acute or chronic infections requiring systemic antibiotic or antiviral therapy at screening.
12. Known human immunodeficiency virus (HIV) infection or positive syphilis test result.
13. Pregnant, lactating, or women planning to become pregnant.
14. Concomitant diseases that may interfere with the conduct of the study, or physical abnormalities that the investigator deems pose an excessive risk to the subject, including but not limited to a history of significant gastrointestinal bleeding within 3 months prior to enrollment or a high risk of bleeding, active peptic ulcer, uncontrolled mental illness, or mental disorders that may interfere with the subject's understanding of the informed consent form or cooperation with treatment.
15. A history of hypersensitivity to ethanol or propylene glycol.
16. Other reasons judged by the investigator that make the subject unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
9-month overall survival rate | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Tianyinshan Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided